CLINICAL TRIAL: NCT01042522
Title: A Randomized Phase II Trial of Paclitaxel and Carboplatin vs. Bleomycin, Etoposide, and Cisplatin for Newly Diagnosed Advanced Stage and Recurrent Chemonaive Sex Cord-Stromal Tumors of the Ovary
Brief Title: Paclitaxel and Carboplatin or Bleomycin Sulfate, Etoposide Phosphate, and Cisplatin in Treating Patients With Advanced or Recurrent Sex Cord-Ovarian Stromal Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0264; NCI-2011-02000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000662814; GOG-0264 (Other: NRG Oncology); GOG-0264 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-01-01; First posted 2010-01-05 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Granulosa Cell Tumor; Ovarian Gynandroblastoma; Ovarian Sertoli-Leydig Cell Tumor; Ovarian Sex Cord Tumor With Annular Tubules; Ovarian Sex Cord-Stromal Tumor; Ovarian Sex Cord-Stromal Tumor, Not Otherwise Specified; Ovarian Steroid Cell Tumor
MeSH Terms: conditions — Granulosa cell tumor of the ovary; Ovarian gynandroblastoma; Sertoli-Leydig Cell Tumor | interventions — Bleomycin; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; etoposide phosphate; Paclitaxel; Taxes

ARMS (2):
- Arm I (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (bleomycin sulfate, etoposide phosphate, cisplatin) (Experimental): Patients receive bleomycin sulfate IV on day 1 and etoposide IV over 1 hour and cisplatin IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cisplatin; Drug: Etoposide Phosphate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bleomycin Sulfate — Given IV
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Bleomycini Sulfas; Blexane; Oil Bleo
  Arms: Arm II (bleomycin sulfate, etoposide phosphate, cisplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (paclitaxel, carboplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm II (bleomycin sulfate, etoposide phosphate, cisplatin)
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
  Arms: Arm II (bleomycin sulfate, etoposide phosphate, cisplatin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (paclitaxel, carboplatin)

SUMMARY:
This randomized phase II trial studies paclitaxel and carboplatin to see how well they work compared with bleomycin sulfate, etoposide phosphate, and cisplatin in treating patients with sex cord-ovarian stromal tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or has returned (recurrent). Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective in treating sex cord-ovarian stromal tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of paclitaxel and carboplatin with respect to progression free survival (using bleomycin, etoposide, and cisplatin [BEP] as a reference) for newly diagnosed advanced or recurrent chemonaive ovarian sex cord-stromal tumors.

SECONDARY OBJECTIVES:

I. To estimate the toxicity of paclitaxel and carboplatin, and bleomycin, etoposide, and cisplatin in this patient population.

II. To estimate overall survival for paclitaxel and carboplatin relative to that of BEP.

III. To evaluate response rate in the subset of patients with measurable disease.

TERTIARY OBJECTIVES:

I. To collect fixed and/or frozen tumor tissue for future translational research studies.

II. To explore the utility of inhibin A and inhibin B as prognostic and predictive biomarkers for ovarian sex cord-stromal tumors and to examine changes in these markers with treatment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bleomycin sulfate IV on day 1 and etoposide phosphate* IV over 1 hour and cisplatin IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who have received prior radiotherapy receive etoposide phosphate on days 1-4.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed ovarian stromal tumor [granulosa cell tumor, ganulosa cell-theca cell tumor, Sertoli-Leydig cell tumor (androblastoma), steroid (lipid) cell tumor, gynandroblastoma, unclassified sex cord-stromal tumor, sex cord tumor with annular tubules]
* Patients must have newly diagnosed, stage IIA - IV disease and must be entered within eight weeks from surgery; they may have either measurable residual disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, or they may have no measurable residual disease; OR, they must have biopsy-proven recurrent disease of any stage and have never received cytotoxic chemotherapy
* Patients must have a Gynecologic Oncology Group (GOG) performance grade of 0, 1, or 2
* Patients of childbearing potential must have a negative serum pregnancy test and must agree to practice an effective means of birth control
* Patients in the measureable disease cohort must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Platelet greater than or equal to 100,000/mcl
* Creatinine no greater than the institutional upper limits of normal
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (CTCAE grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3.0 x ULN (CTCAE grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE grade 1
* No signs of clinically significant hearing loss
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have pulmonary function sufficient to receive bleomycin, with normal lung expansion, absence of crackles on auscultation, and normal carbon monoxide diffusion (DLCO), defined as greater than 80% predicted
* Patients with a history of hypersensitivity reactions to prior chemotherapy administered for previous cancer diagnoses are eligible to participate in the study, unless the hypersensitivity reaction consisted of anaphylaxis not amenable to desensitization
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients must be entered within 8 weeks after surgery performed for either 1) initial diagnosis, staging, and/or cytoreduction, or 2) (if done) management of recurrent disease in a chemonaive patient
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted

Exclusion Criteria:

* Patients who have received any prior cytotoxic chemotherapy or biologics for sex cord-stromal tumors (SCSTs)
* Patients with apparent stage I disease who have not undergone a staging procedure
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years
* Woman who are pregnant or breastfeeding
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator can consult the study chair or study co-chairs for uncertainty in this regard

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2022-11-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jubilee Brown, Principal Investigator — NRG Oncology
Locations (219):
- United States (219):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Brown J, Miller A, Holman LL, Backes F, Nagel C, Bender D, Miller DS, Powell MA, Westin SN, Bonebrake A, Muller CY, Secord AA, Crane E, Schorge J, Tew WP, Sood AK, Bookman MA, Aghajanian C, Gershenson DM. Results of a randomized phase II trial of paclitaxel and carboplatin versus bleomycin, etoposide and cisplatin for newly diagnosed and recurrent Chemonaive stromal ovarian tumors: An NRG oncology/gynecologic oncology group study14. Gynecol Oncol. 2024 Nov;190:283-290. doi: 10.1016/j.ygyno.2024.09.002. Epub 2024 Sep 12. PMID 39265466

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin)
Started | 31 | 32
Completed | 23 (Completed 6 cycles of protocol regimen) | 26 (Completed 4 cycles of protocol regimen)
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Disease Progression | 5 | 0
Not completed — Death | 1 | 0
Not completed — Patient Refused | 0 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin) | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.71 (12.51) | 44.05 (13.86) | 47.33 (13.53)
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 years | 2 | 7 | 9
  30 - 39 years | 2 | 5 | 7
  40 - 49 years | 13 | 6 | 19
  50 - 59 years | 6 | 10 | 16
  >= 60 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Performance Status [Count of Participants; unit: Participants] — For Performance Status, the GOG- score was used:
  0 = normal activity, asymptomatic
  1. = symptomatic, fully ambulatory
  2. = symptomatic, in bed < 50% of time
  3. = symptomatic, in bed > 50% of time
  4. = 100% bedridden
  Participants
    0 | 21 | 28 | 49
    1 | 9 | 4 | 13
    2 | 1 | 0 | 1
Measurable Disease [Count of Participants; unit: Participants]
  Measurable Disease | 11 | 12 | 23
  No Measurable Disease | 20 | 20 | 40
Cell Type [Count of Participants; unit: Participants]
  Lipid Cell Tumor | 1 | 0 | 1
  Granulosa Cell Tumor | 28 | 27 | 55
  Sex Cord Stromal Tumor, Unclassified | 2 | 2 | 4
  Sertoli-leydig Cell Tumor | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The relationship of randomized treatment to progression free survival. The RECIST 1.1 criteria are used for disease progression. This is the criteria: progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From start of treatment to time of progression or death, whichever occurs first. Median follow-up time was 48 months.
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin)
Number analyzed (Participants) | 31 | 32
months | 27.7 [11.2 to 41.0] | 19.7 [10.4 to 52.7]

2. Secondary Outcome: Tumor Response Rate
Description: Proportion of evaluable patients with complete or partial tumor response by RECIST 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. (ORR = CR + PR).
Time Frame: Median followup time was 48 months.
Population: Patients with at least one target lesion by RECIST 1.1 criteria and and at least one CT tumor assessment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin)
Number analyzed (Participants) | 14 | 13
proportion of participants | 0.43 [0.21 to 0.67] | 0.54 [0.29 to 0.77]

3. Secondary Outcome: Overall Survival (OS)
Description: The relationship of treatment to overall survival will be assessed. The number of death events in the treatment arm is reported.
Time Frame: From start of treatment to time of death or the date of last contact, assessed up to 10 years. Median follow-up time was 48 months.
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin)
Number analyzed (Participants) | 31 | 32
Participants | 5 | 8

4. Other Pre Specified Outcome: Change in Inhibin A and Inhibin B Levels
Description: Pre-treatment levels of inhibin A and inhibin B will be examined in relation to OS and PFS in Cox proportional hazards models. Changes from baseline in inhibin levels will be compared between treatment groups using mixed effects models accounting for the longitudinal nature of the data. The repeated measures of inhibin will also be explored versus overall survival and PFS using time-dependent covariates in Cox proportional hazards models.
Time Frame: Baseline to up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse events were assessed during the treatment period and up to 100 days after stopping study treatment (an average of 33 months).
Arm/Group | Arm I (Paclitaxel, Carboplatin) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin)
All-Cause Mortality (participants affected / at risk) | 5/31 | 8/32
Serious Adverse Events (participants affected / at risk) | 6/31 | 11/32
Other Adverse Events (participants affected / at risk) | 31/31 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin) (N=31) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin) (N=32)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Death Nos (General disorders) | 1 | 0
Neutrophil Count Decreased (Investigations) | 5 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin) (N=31) | Arm II (Bleomycin Sulfate, Etoposide Phosphate, Cisplatin) (N=32)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 26 | 26
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 4
Cardiac Disorders - Other (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 3 | 11
Ear Pain (Ear and labyrinth disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Endocrine Disorders - Other (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 2 | 0
Watering Eyes (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 18 | 11
Diarrhea (Gastrointestinal disorders) | 7 | 9
Vomiting (Gastrointestinal disorders) | 9 | 14
Abdominal Pain (Gastrointestinal disorders) | 5 | 11
Mucositis Oral (Gastrointestinal disorders) | 3 | 8
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 22 | 25
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Esophageal Pain (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
General Disorders And Administration Site Conditions (General disorders) | 0 | 4
Pain (General disorders) | 8 | 4
Neck Edema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Injection Site Reaction (General disorders) | 1 | 0
Flu Like Symptoms (General disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 2
Edema Limbs (General disorders) | 3 | 7
Fatigue (General disorders) | 23 | 23
Fever (General disorders) | 4 | 4
Chills (General disorders) | 1 | 2
Infusion Related Reaction (General disorders) | 2 | 3
Allergic Reaction (Immune system disorders) | 1 | 1
Wound Infection (Infections and infestations) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 3 | 1
Papulopustular Rash (Infections and infestations) | 1 | 0
Mucosal Infection (Infections and infestations) | 0 | 2
Lung Infection (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0
Vaginal Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 3
Catheter Related Infection (Infections and infestations) | 0 | 1
Bronchial Infection (Infections and infestations) | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Investigations - Other (Investigations) | 1 | 2
Weight Loss (Investigations) | 1 | 2
Weight Gain (Investigations) | 1 | 4
Platelet Count Decreased (Investigations) | 17 | 15
Lymphocyte Count Decreased (Investigations) | 0 | 6
Ggt Increased (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 1 | 1
Cholesterol High (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 26 | 29
Carbon Monoxide Diffusing Capacity Decreased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 22 | 27
Aspartate Aminotransferase Increased (Investigations) | 4 | 1
Alkaline Phosphatase Increased (Investigations) | 3 | 4
Alanine Aminotransferase Increased (Investigations) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 6
Hypokalemia (Metabolism and nutrition disorders) | 1 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 10 | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal And Connective Tissue Disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 19 | 13
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 7 | 12
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 6
Cognitive Disturbance (Nervous system disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 6
Depression (Psychiatric disorders) | 4 | 7
Confusion (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 5 | 6
Urinary Urgency (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Urinary Tract Pain (Renal and urinary disorders) | 1 | 4
Urinary Frequency (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 3
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 2 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Respiratory, Thoracic And Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 3
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 19
Thromboembolic Event (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 6 | 5
Hot Flashes (Vascular disorders) | 8 | 6
Hematoma (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
An interim analysis was planned occur after 20 PFS events were observed in either arm (roughly 50% information time). The futility threshold for paclitaxel and carboplatin relative to BEP was HR>1.10. Median followup time was 48 months.

The study closed at the interim analysis for futility, and difficulty with accrual. At the time of closures, 63 of a planned 128 patients had enrolled at the time of accrual suspension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT01042522/Prot_SAP_000.pdf